CLINICAL TRIAL: NCT05682950
Title: A Prospective Study to Evaluate Optimal Margin of Iterative Cone-beam Computed Tomography Guided Online Adaptive Radiotherapy for Postoperative Treatment of Endometrial and Cervical Cancer
Brief Title: Optimal Margin Evaluation of Online Adaptive Radiotherapy for Postoperative Treatment of Endometrial and Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-ART
Record Dates: First submitted 2022-12-14; First posted 2023-01-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Uterine Cervical Neoplasm; Endometrial Neoplasms
Keywords: Uterine Cervical Neoplasm; Endometrial Neoplasms; Online Adaptive Radiotherapy; Adjuvant Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online Adaptive Radiotherapy (Experimental): Patients receive online adaptive radiotherapy. The CTV contours of the following areas: vaginal cuff, obturator nodal chain, internal iliac nodal chain, external iliac nodal chain, presacral nodal chain and common iliac nodal chain. The upper border of CTV is at the level of aortic bifurcation. A dose of 45-50.4Gy is delivered to CTV with online adaptive radiotherapy.
  Interventions: Radiation: online adaptive radiotherapy

INTERVENTIONS:
Radiation: online adaptive radiotherapy — CTV covers pelvis.

SUMMARY:
Online adaptive radiotherapy has demonstrated to be feasible to reduce inter-fractional radiotherapy errors as it re-optimizes treatment plan every fraction. To investigate the extent and value of margin reduction，we conduct a prospective clinical trial to determine the optimal margin and toxicity of smaller margin.

DETAILED DESCRIPTION:
This is a prospective phase II clinical trial with an anticipated total of more than 380 radiotherapy fractions of 15 patients to evaluate optimal margin of iterative cone-beam computed tomography（iCBCT） guided online adaptive radiotherapy （oART） for postoperative treatment of endometrial and cervical cancer. Postoperative endometrial and cervical cancer patients with following characteristics are included in the present study:（a）underwent radical surgery （b）no residual tumor at the resection margin by postoperative pathology（c）pathological findings indicate risk factors but no metastasis (d) adjuvant radiotherapy are prescribe (e)without evidence of para-aortic metastatic lymph nodes. Five patients （almost 125 fractions）treated with oART have the target volume contoured on pre-treatment iCBCTs and end-treatment iCBCTs. Anterior-posterior, lateral, and superior-inferior shifts were calculated and the average shift in all directions was calculated. A clinical target volume (CTV) to planing tumor volume (PTV) expansion is determined and verifies on a validation cohort of 10 patients (almost 250 fractions) treated with oART. Record acute toxicity from the start of treatment to 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent before treatment.
2. Postoperative endometrial and cervical cancer patients with pathologically confirmed no residual tumor at the resection margin and no evidence of distant metastasis (FIGO stage IVB).
3. Pathological findings indicate risk factors and adjuvant radiotherapy are prescribe.
4. Karnofsky score ≥ 70.
5. Subjects aged ≥ 18 years and ≤ 70 years.
6. No evidence of para-aortic metastatic lymph nodes.
7. No contraindications to CT scanning.
8. Subjects must be able to cooperate in completing the entire study.
9. Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L.
10. Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

Exclusion Criteria:

1. Subjects who have received prior pelvic radiotherapy.
2. Subjects with other primary malignancies.
3. Subjects with contraindications to radiotherapy, as determined by the investigators.
4. Any severe disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.
5. Active infection with fever.
6. Active inflammatory bowel disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The dose coverage of target volume as assessed by planing tumor volume V100% | Through study completion, total an average of six month
  Planing tumor volume V100%, defined as the planing tumor volume receiving at least 100% of the prescribed dose (V100%), is used to evaluate the dose coverage of target volume.
A minimum PTV margin could encompass CTV | Through study completion, toral an average of six month
  Expansions were applied to the pretreatment PTV to assess required minimum margin required to encompass the postreatment CTV.

SECONDARY OUTCOMES:
Safety for treatment as assessed by organs at risk doses | Through study completion, total an average of six month
  Safety for treatment was mainly evaluated by the organs at risk doses, including bladder, rectum, bone marrow, etc
Number of participants with acute toxicity as assessed by CTCAE 5.0 | From the start of treatment to 3 months after treatment
  Evaluated with CTCAE 5.0
Adaptive time data | Through study completion, total an average of six month
  For each treatment in each fraction, adaptive time was recorded from first cone beam computed tomography (CBCT) to the selection of the preferred plan for the treatment.
Target contouring accuracy | Through study completion, total an average of six month
  For every target in each fraction, the evaluation of accuracy for target contouring are categorized as follow: no edits, minor edits, moderate edits, major edits and not applicable.
Organs at risk contouring accuracy | Through study completion, total an average of six month
  For every organs at risk in each fraction, the evaluation of accuracy for organs at risk contouring are categorized as follows: no edits, minor edits, moderate edits, major edits and not applicable.
Late toxicity evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme | total an average of 2-year
  Evaluated every three months with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Zhang, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jong R, Visser J, van Wieringen N, Wiersma J, Geijsen D, Bel A. Feasibility of Conebeam CT-based online adaptive radiotherapy for neoadjuvant treatment of rectal cancer. Radiat Oncol. 2021 Jul 23;16(1):136. doi: 10.1186/s13014-021-01866-7. PMID 34301300
- [Background] Schiff JP, Stowe HB, Price A, Laugeman E, Hatscher C, Hugo GD, Badiyan SN, Kim H, Robinson CG, Henke LE. In Silico Trial of Computed Tomography-Guided Stereotactic Adaptive Radiation Therapy (CT-STAR) for the Treatment of Abdominal Oligometastases. Int J Radiat Oncol Biol Phys. 2022 Dec 1;114(5):1022-1031. doi: 10.1016/j.ijrobp.2022.06.078. Epub 2022 Jun 26. PMID 35768023